CLINICAL TRIAL: NCT00967967
Title: Validation of a Rhinitis Control Tool : the Rhinitis Control Scoring System (RCSS)
Brief Title: Validation of the Rhinitis Control Scoring System (RCSS)
Acronym: RCSS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting results from sub analysis to decide if study continuesé
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, Professeur, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER 20389
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Asthma; Rhinitis
Keywords: control; symptoms
MeSH Terms: conditions — Asthma; Rhinitis | interventions — desloratadine; Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mometasone furoate and desloratadine (Other): Mometasone and desloratadine treatment
  Interventions: Drug: Medication Mometasone furoate and desloratadine

INTERVENTIONS:
Drug: Medication Mometasone furoate and desloratadine — One month treatment with both drugs
  Other Names: Nasonex; Aerius

SUMMARY:
Many patients suffering from allergic rhinitis do not recognize or perceive their symptoms. Instruments have been developed to assess quality of life in rhinitis, asthma or both, but there is a need to develop validated tools or methods to assess rhinitis control among rhinitis and/or asthmatic patients. The aim of this study is to assess the discriminative and evaluative properties of the RCSS in asthmatic patients with allergic rhinitis.

DETAILED DESCRIPTION:
Allergic asthmatic subjects showing seasonal rhinitis symptoms will be recruited. The discriminative (internal consistency, cross sectional construct validity and reliability) and evaluative (responsiveness and longitudinal construct validity) properties of the RCSS will be evaluated as well as the relationship between rhinitis control and asthma control. RCSS will be completed at various time points during the seasonal allergic period.

ELIGIBILITY:
Inclusion Criteria:

* asthma
* seasonal allergic rhinitis

Exclusion Criteria:

* smoking
* nasal polyposis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Discriminative (internal consistency, cross sectional construct validity and reliability) and evaluative (responsiveness and longitudinal construct validity) properties of the RCSS. | March to November 2009

SECONDARY OUTCOMES:
The relationship between rhinitis control and asthma control. | March to November 2009

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Boulay ME, Boulet LP. The Rhinitis Control Scoring System: Development and validation. Am J Rhinol Allergy. 2016 Jan-Feb;30(1):54-9. doi: 10.2500/ajra.2016.30.4260. PMID 26867531